CLINICAL TRIAL: NCT02744950
Title: A Prospective, Randomized Study to Evaluate the Efficacy of Pulley Closures Compared to Intermediate or Complex Closures for Reconstruction of Scalp Surgical Defects
Brief Title: Comparison of Scar Results and Time for Closures of Scalp Defects Via Pulley Sutures or Layered Repairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Dermatologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SK1234
Record Dates: First submitted 2016-04-14; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Scar
Keywords: pulley; scalp defects
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermediate/complex repair (Active Comparator): This arm will have closures of scalp defects with deep and superficial suture placement.
  Interventions: Procedure: Intermediate Repair
- Pulley stitches (Experimental): This arm of the study will have only pulley stitches to close the entire defect.
  Interventions: Procedure: Pulley stitches

INTERVENTIONS:
Procedure: Pulley stitches
  Arms: Pulley stitches
Procedure: Intermediate Repair
  Arms: Intermediate/complex repair

SUMMARY:
Surgical defects on the scalp require closure via various techniques of suture placement. A traditional technique requires both dermal (deep) and epidermal (superficial) placement of sutures to close the defect; this is referred to as intermediate or complex linear repair. However, the scalp is a location with high tension, and thus the closures take an hour or longer to perform. A type of suture placement referred to as the "pulley stitch" requires placement of a few stitches along the defect. The pulley stitch can be used in areas of high tension to close a large defect. The purpose of this study is to compare the scar results and time taken to perform scalp closures via only pulley stitches or via intermediate/complex linear repairs.

To my knowledge, no such study has been performed to compare the two techniques. Such a study would be useful in demonstrating comparable scar appearance and reduce the time to perform scalp closures.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Ability to understand risks, benefits, and alternatives to the study and to be able to give an informed consent
3. Lesions such as skin cancer or benign lesions on the scalp amenable to surgical excision or to MOHS surgical technique
4. Frontal scalp defects defined as frontal hair line to crown of scalp
5. Scalp defect size of 2cm - 8 cm

Exclusion criteria:

1. Patients who tend to form keloids or hypertrophic scars
2. Patients with a history of scleroderma or morphea
3. Pregnant or breast-feeding females
4. Patients whose surgical defects require flap closures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to close wound | Depends on case typically 4-10 minutes
  Time it takes to close the defect in each arm; measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System- Dermatology, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Via a research paper